CLINICAL TRIAL: NCT05547828
Title: Safety and Efficacy of Tislelizumab Combined With Chemoradiotherapy in First-line Treatment of Stage IVb Esophageal Squamous Cell Carcinoma
Brief Title: Efficacy and Safety of Tislelizumab and Nab-paclitaxel Combined With Low-dose Radiotherapy in Patients With Stage IVb Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD-CR-ESCC
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: ESCC
Keywords: PD-1; RCT; Ⅳb ESCC; 1 line
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Masking Description: This study is a single-arm, prospective, open-label clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with chemoradiotherapy (Other): Tislelizumab: According to the instructions of tislelizumab, 200 mg intravenously on the first day of each cycle, 21 days as a cycle.
  Nab-paclitaxel: white purple: 100mg/m2 intravenous infusion on d1.8.15 (during chemotherapy) 100mg/m2 intravenous infusion q3w ╳ 3 cycles (during consolidation therapy) Radiotherapy: 40Gy/20f, 5 times/w, (esophageal primary tumor and metastatic lymph nodes)
  Interventions: Drug: Tislelizumab combined with chemoradiotherapy

INTERVENTIONS:
Drug: Tislelizumab combined with chemoradiotherapy — Tislelizumab: According to the instructions of tislelizumab, 200 mg intravenously on the first day of each cycle, 21 days as a cycle.
  Nab-paclitaxel: white purple: 100mg/m2 intravenous infusion on d1.8.15 (during chemotherapy) 100mg/m2 intravenous infusion q3w ╳ 3 cycles (during consolidation therapy) Radiotherapy: 40Gy/20f, 5 times/w, (esophageal primary tumor and metastatic lymph nodes)

SUMMARY:
This study is a single-arm, prospective, open-label clinical study to evaluate the safety and efficacy of tislelizumab combined with chemoradiotherapy in first-line treatment of patients with stage IVb esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study is a single-center, prospective, single-arm, open-label study. It will explore the efficacy and safety of tislelizumab combined with nab-paclitaxel in the first-line treatment of stage IVb esophageal squamous cell carcinoma on the basis of low-dose radiotherapy（40Gy/20f，5次/w）. To explore new treatment modalities and prolong patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of Esophageal squamous cell carcinoma

   -diagnosed with stage IVb Esophageal squamous cell carcinoma (UICC/AJCC 8th edition TNM staging system) by CT/MRI/PET-CT/ECT, laboratory examination and pathological examination results; specific: any T, any N, M1;
2. No previous anti-tumor treatment; expected survival period of more than half a year; 3.18-75 years old, PS score 0-1;

4. According to RECIST1.1 criteria, there is at least one measurable target lesion, and tumor imaging evaluation is performed within 28 days before the first dose; 5. Major organ function is normal, that is, the following criteria are met: 6. No active autoimmune disease; 7. No active hepatitis; 8. General conditions or medical complications can tolerate radiotherapy, chemotherapy and immunotherapy; 9. No history of malignant tumor, no previous anti-tumor therapy; 10. For premenopausal or surgically sterilized female patients: Consent to abstinence or use of effective contraception during treatment and for at least 7 months after the last dose of study treatment; 11. Understand and sign the informed consent form for this study.

Exclusion Criteria:

1. Previous antitumor therapy or radiation therapy for any malignant tumor;
2. patients receiving standard treatment;
3. concurrently receiving anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy, or immunotherapy;
4. Has undergone major surgical procedures unrelated to colorectal cancer within 4 weeks prior to enrollment, or the patient has not fully recovered from such surgical procedures;
5. Serious heart disease or discomfort, including but not limited to the following:
6. Inability to swallow, bowel obstruction, or other factors that interfere with drug taking and absorption;
7. Known history of allergy to the drug components of this regimen; history of immunodeficiency, including positive HIV test, positive HBV/HCV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
8. Pregnant or lactating female patients, female patients of childbearing potential with a positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial period and within 7 months after the last study drug;
9. Have serious comorbidities or other comorbidities that would interfere with planned treatment, or any other condition that the investigator considers the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  It is defined as the number of subjects with the best response effect as complete remission (CR) or partial remission (PR) during the period from the start of the subjects receiving the treatment regimen of this study to the progression of the subjects' disease in the total number of subjects in the analysis data set. percentage of the population（%）.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 24 months
  Defined as the number of subjects whose tumors shrank or remained stable for a certain period of time from receiving the treatment regimen of this study to the progression of the subject's disease, including complete remission (CR) and partial remission (PR) in the analysis data set percentage of the total population（%）.
Progression Free Survival (PFS) | Up to 24 months
  Defined as the time from randomization to tumor progression in any aspect or death from any cause（Unit: month）.
  Assessed according to RECIST 1.1 criteria, analysis of this indicator included tumor evaluation results during study treatment and follow-up. If the patient has several indicators that can be judged as PD, the first indicator will be used for PFS analysis; recurrence, new lesions or death are considered to have reached the end of the study, and the patient is treated with other systemic or target-targeted anti-PD. Tumor treatment is also considered tumor progression.
Overall survival (OS) | Up to 24 months
  Defined as the time from randomization to death from any cause（Unit: month）.
Drug-Related Safety Indicators | Up to 24 months
  Exposure to the investigational drug and incidence, nature, and severity of adverse events, including serious adverse events（n，%）。